CLINICAL TRIAL: NCT02681198
Title: Lofexidine Pharmacokinetics in the Presence of Paroxetine, a Strong CYP2D6 Inhibitor, in Healthy Volunteers
Brief Title: Lofexidine Pharmacokinetics in the Presence of Paroxetine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM-LX1-1010; U01DA033276 (NIH)
Record Dates: First submitted 2016-02-01; First posted 2016-02-12 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Healthy; Lofexidine; Paroxetine; Volunteer
MeSH Terms: interventions — lofexidine; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lofexidine and paroxetine (Experimental): Lofexidine in the presence of paroxetine
  Interventions: Drug: Lofexidine; Drug: Paroxetine

INTERVENTIONS:
Drug: Lofexidine — All subjects will receive two single doses of lofexidine HCl; one 0.4 mg dose taken alone on Day 1 and one 0.4 mg dose taken with 40 mg once daily paroxetine HCl at steady-state on Day 13.
Drug: Paroxetine — All subjects will receive daily single doses of paroxetine HCl; one 20 mg dose taken Days 4-6, one 40 mg dose taken Days 7-19, one 20 mg dose taken Day 20, one 10 mg dose taken Days 21-22.

SUMMARY:
The purpose of this study is to determine the pharmacokinetics, safety and tolerability of lofexidine HCl in the presence of paroxetine in healthy adults.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-sequence study to determine the pharmacokinetics, safety and tolerability of lofexidine HCl in the presence of paroxetine in healthy adults. Lofexidine HCl is an alpha-2 adrenergic agonist under development for the treatment of acute withdrawal from short-acting opioids. Paroxetine HCl is an orally administered psychotropic drug indicated in the treatment of major depressive, obsessive compulsive, panic, social anxiety, and generalized anxiety disorders. Paroxetine is a strong CYP2D6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between ages of 18 to 60 years at enrollment with a body mass index (BMI) between 18 and 35 kg/m2.
* Female subjects must not be lactating, and must either a) be postmenopausal or b) agree to use an acceptable form of birth control from screening until 14 days after completion of the study.
* Subject is in good health based on medical history, physical exam, laboratory profile, and electrocardiogram (ECG) as judged by the Investigator.
* If subject smokes, subject agrees to limit smoking while in the study to not more than 10 cigarettes per day.

Exclusion Criteria:

* History of suicidal ideations or depression requiring professional intervention including counseling or antidepressant medication over the past 12 months.
* History or presence of allergic or adverse response to lofexidine, paroxetine, or related drugs.
* Received any drugs capable of inhibiting CYP enzymes CYP1A2, CYP2C19, or CYP2D6 within 14 days or 5 half-lives (whichever is more) before Day 1.
* Consumes more than 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) or has a significant history of alcohol abuse or drug/chemical abuse within the last 1 year.
* Has a history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0 hour (predose) and 0.25, 0.5, 1, 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48 and 72 hours after lofexidine Dose 1; 0 hour (predose) and 0.25, 0.5, 1 , 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48, 72, 96, 120, 144 and 168 hours after lofexidine Dose 2.
Time to Maximum Plasma Concentration (Tmax) | 0 hour (predose) and 0.25, 0.5, 1, 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48 and 72 hours after lofexidine Dose 1; 0 hour (predose) and 0.25, 0.5, 1 , 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48, 72, 96, 120, 144 and 168 hours after lofexidine Dose 2.
Apparent Terminal Elimination Half-life (T½) | 0 hour (predose) and 0.25, 0.5, 1, 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48 and 72 hours after lofexidine Dose 1; 0 hour (predose) and 0.25, 0.5, 1 , 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48, 72, 96, 120, 144 and 168 hours after lofexidine Dose 2.
Area Under the Concentration-Time Curve from Time Zero to Last Quantified Concentration (AUC 0-t) | 0 hour (predose) and 0.25, 0.5, 1, 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48 and 72 hours after lofexidine Dose 1; 0 hour (predose) and 0.25, 0.5, 1 , 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48, 72, 96, 120, 144 and 168 hours after lofexidine Dose 2.
Area Under the Curve from Time Zero to Infinity (AUC 0-infinity) | 0 hour (predose) and 0.25, 0.5, 1, 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48 and 72 hours after lofexidine Dose 1; 0 hour (predose) and 0.25, 0.5, 1 , 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48, 72, 96, 120, 144 and 168 hours after lofexidine Dose 2.
Apparent Clearance (CL/F) | 0 hour (predose) and 0.25, 0.5, 1, 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48 and 72 hours after lofexidine Dose 1; 0 hour (predose) and 0.25, 0.5, 1 , 2, 3, 4, 5, 6.5, 8, 12, 16, 24, 32, 48, 72, 96, 120, 144 and 168 hours after lofexidine Dose 2.

SECONDARY OUTCOMES:
Blood pressure (sitting and standing) | screening; predose and 3.5 and 7.5 hours postdose on Days 1, 13; Day 22.
Heart rate (sitting and standing) | screening; predose and 3.5 and 7.5 hours postdose on Days 1 and 13; Day 22.
Laboratory Assessments | screening; Day -1, 2, 12, 14; Day 22.
  Measurements in hematology, blood chemistry, coagulation, and urinalysis parameters will be examined. Labs will be done at screening, and at Days -1, 2,12,14, 22.
12-lead ECGs | screening; 0 and 6.5 hours postdose on Days 1, 12, 13; Day 22.
Holter ECGs | 0 (predose), and 3, 4 and 8 hours postdose on Days 1, 12, 13
Columbia Suicide Severity Rating Scale (C-SSRS) | screening; Days 7, 13, 22, 50.

CONTACTS AND LOCATIONS:
Overall Officials: George J Atiee, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No